CLINICAL TRIAL: NCT01178216
Title: Use of Immune Globulin Intravenous (Human), 10% (IVIG), Plus Rituximab as Agents to Reduce Donor Specific Antibodies, Improve Transplant Rates and Outcomes in Highly-HLA Sensitized Patients Awaiting Deceased Donor Kidney Transplantation
Brief Title: Use of Immune Globulin Plus Rituximab for Desensitization in Highly HLA Sensitized Patients Awaiting Deceased Donor Kidney Transplantation
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Stanley Jordan, MD (Other)
Collaborators: Genentech, Inc. (Industry)
Responsible Party: Sponsor-Investigator, Stanley Jordan, MD, Medical Director, Medical Director, Renal Transplantation & Transplant Immunotherpay, Cedars-Sinai Medical Center
Organization: Cedars-Sinai Medical Center (Other)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: Genentech-Ritux2010
Record Dates: First submitted 2010-08-09; First posted 2010-08-10 (Estimated); Results first posted 2018-09-07 (Actual); Last update posted 2018-10-26 (Actual); Status verified 2018-09

CONDITIONS: End Stage Renal Disease
Keywords: Kidney transplant; highly sensitized
MeSH Terms: conditions — Kidney Failure, Chronic | interventions — Rituximab

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Rituxan (Experimental): All study patients will receive Rituxan 1g on day 15 from start of desensitization and either 3M or 6M post transplant depending on the presence of DSA.
  Interventions: Biological: Rituxan

INTERVENTIONS:
Biological: Rituxan — Rituximab (1gm) given on day# 15. Transplanted patients will receive an additional dose of Rituximab at 3M if DSA remains or 6M if denovo DSA present.
  Other Names: Rituximab

SUMMARY:
This single center, Phase I/II, exploratory study has been modified to a safety/efficacy study providing all patients with IVIG and Rituximab. The trial will examine the safety and efficacy of human polyclonal IVIG 10%, when given at [2.0 gm/kgx2], + Rituximab 1gm to reduce donor-specific antibodies (DSA) to a level that is permissive for transplantation in 75 subjects (adults only ages >18 yrs) who are highly-HLA sensitized and are awaiting deceased donor kidney transplant. Once transplant offers are entertained, a donor-specific crossmatch will be performed. If acceptable crossmatches and DSA levels are seen, the patients will proceed to DD transplantation. Patients receiving transplants will receive an additional dose of IVIG at transplantation (within 10 days) and will receive additional doses of Rituximab 1g at 3M post transplant if DSA levels remain or become positive at 6M if de novo DSA occur. Patients who are desensitized and not transplanted at 9M after desensitization will have completed the study and can be treated as best judged by their physician.

DETAILED DESCRIPTION:
Organ transplantation offers the only hope for a normal life for patients with end-stage renal disease on dialysis. For patients with antibodies to human leukocyte antigens (HLA), transplantation is extremely difficult or impossible since pre-formed antibodies will cause severe rejection and loss of transplanted organs. Intravenous gamma globulin (IVIG) can reduce or eliminate these antibodies in most patients and allow for successful transplantation. This breakthrough has allowed patients previously considered not transplantable to receive life-saving transplants. However, IVIG alone does not always eradicate the anti-HLA antibodies to a degree that will allow transplantation.

In this study, the investigators propose additional treatment with rituximab, a humanized antibody directed at the CD20 antigen that is present on most B-cells. Both IVIG and rituximab are approved by the U.S. Food and Drug Administration (FDA) for numerous immunologic disorders and Non-Hodgkin's lymphoma, respectively. However, neither is approved by the FDA for desensitization of highly-HLA sensitized transplant patients. A previously conducted pilot study demonstrated IVIG + Rituximab can fill an important gap in the current therapeutic approach for management of highly sensitized patients and may become the standard therapy.

Update: Study updated after observation that subjects transplanted after desensitization with IVIG alone experienced higher rates of antibody rejection and graft loss. The primary objective of this revised protocol will be to examine the safety and efficacy of IVIG 2gm/kg (maximum 140g) given on day#0 & day #30 plus Rituximab 1gm given on day #15. Transplanted patients will receive additional doses of Rituximab 1gm at 3 months post-transplant if donor specific antibody (DSA) levels remain or become positive or at 6M if de novo DSA occur. All transplanted patients who remain DSA negative, will not receive additional Rituximab. All transplanted patients will have a protocol biopsy at transplant and 12 months. All subjects will complete 5 visits in the pre-transplant phase of the study. Patients who are transplanted will have additional 5 post-transplant visits. The following are research-related procedures:

1. Rituximab infusion.
2. Kidney allograft biopsies (Intra-op, 12 months post-transplant)
3. Rituximab level, HACA levels
4. Immunologic biomarkers (CD19+, CD38+, CD27+)

Although the investigator commonly uses both treatment regimens at Cedars-Sinai Medical Center, only the IVIG treatment is considered to be standard of care for highly HLA-sensitized patients. The investigational component of this study is the addition of the rituximab. Currently the study has been amended to a safety and efficacy study focusing on decreasing HLA antibodies pre-transplant and minimizing DSA post-transplant.

ELIGIBILITY:
Inclusion Criteria:

1. End-stage renal disease.
2. No known contraindications for therapy with IGIV10%/Rituximab.
3. Age 18-70 years at the time of screening.
4. PRA> 30% demonstrated on 3 consecutive samples, UNOS wait time sufficient to allow DD offers, history of sensitizing events, positive crossmatch with the intended donor.
5. Subject/Parent/Guardian must be able to understand and provide informed consent.

Exclusion Criteria:

1. Lactating or pregnant females.
2. Pediatric patients <18 years of age
3. Women of child-bearing age who are not willing or able to practice FDA-approved forms of contraception.
4. HIV-positive subjects.
5. Subjects who test positive for HBV infection [positive HBVsAg, HBVcAg, or HBVeAg/DNA] or HCV infection [positive Anti-HCV (EIA) and confirmatory HCV RIBA].
6. Subjects with active TB.
7. Subjects with selective IgA deficiency, those who have known anti-IgA antibodies, and those with a history of anaphylaxis or severe systemic responses to any part of the clinical trial material.
8. Subjects who have received or for whom multiple organ transplants are planned.
9. Recent recipients of any licensed or investigational live attenuated vaccine(s) within two months of the screening visit (including but not limited to any of the following:

   * Adenovirus [Adenovirus vaccine live oral type 7]
   * Varicella [Varivax]
   * Hepatitis A [VAQTA]
   * Rotavirus [Rotashield]
   * Yellow fever [Y-F-Vax]
   * Measles and mumps [Measles and mumps virus vaccine live]
   * Measles, mumps, and rubella vaccine [M-M-R-II]
   * Sabin oral polio vaccine
   * Rabies vaccines [IMOVAX Rabies I.D., RabAvert])
10. A significantly abnormal general serum screening lab result defined as a WBC < 3.0 X 103/ml, a Hgb < 8.0 g/dL, a platelet count < 100 X 103/ml, , an SGOT > 5X upper limit of normal, and an SGPT >5X upper limit of normal range.
11. Individuals deemed unable to comply with the protocol.
12. Subjects with active CMV or EBV infection as defined by CMV-specific serology (IgG or IgM) and confirmed by quantitative PCR with or without a compatible illness.
13. Subjects with a known history of previous myocardial infarction within one year of screening.
14. Subjects with a history of clinically significant thrombotic episodes, and subjects with active peripheral vascular disease.
15. Use of investigational agents within 4 weeks of participation.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 41 (Actual)
Dates: Start 2013-09; Primary Completion 2017-07-28 (Actual); Study Completion 2017-07-28 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Stanley Jordan, MD, Principal Investigator — Cedars-Sinai Medical Center
Locations (1):
- Cedars-Sinai Medical Center, Los Angeles, California, United States

REFERENCES:
- [Background] Jordan SC, Peng A, Vo AA. Therapeutic strategies in management of the highly HLA-sensitized and ABO-incompatible transplant recipients. Contrib Nephrol. 2009;162:13-26. doi: 10.1159/000170864. Epub 2008 Oct 31. PMID 19001810
- [Background] Vo AA, Lukovsky M, Toyoda M, Wang J, Reinsmoen NL, Lai CH, Peng A, Villicana R, Jordan SC. Rituximab and intravenous immune globulin for desensitization during renal transplantation. N Engl J Med. 2008 Jul 17;359(3):242-51. doi: 10.1056/NEJMoa0707894. PMID 18635429
- See also: Cedars-Sinai Medical Center Kidney Transplant Website — http://www.cedars-sinai.edu/Patients/Quality-Measures/Clinical-Areas/Transplantation/Kidney-Transplantation.aspx

RESULTS

PARTICIPANT FLOW:
Recruitment Details: From 2013 - 2017, Highly Sensitized (HS) patients with calculated panel reactive antibodies (CPRA)>50% underwent desensitization while awaiting kidney transplantation
Period: Overall Study
Arm/Group | Rituxan
Started | 41
Completed | 39
Not Completed | 2

BASELINE CHARACTERISTICS:
Population: From 2013 - 2017, Highly Sensitized (HS) patients with calculated panel reactive antibodies (CPRA)>50% underwent desensitization while awaiting kidney transplantation
Arm/Group | Rituxan
Number analyzed (Participants) | 41
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 40
  >=65 years | 1
Age, Continuous [Median (Inter-Quartile Range); unit: years] | 48 [23 to 69]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 16
  Male | 25
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 0
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 6
  White | 0
  More than one race | 0
  Unknown or Not Reported | 35
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 41

OUTCOME MEASURES:

1. Primary Outcome: Number of Patients That Underwent Transplantation
Description: This trial is designed to determine if Rituximab + IVIG can improve rates of transplantation for highly-HLA sensitized DD candidates on the UNOS waiting list over a 9M period of time after completion of treatment.
Time Frame: 9 month
Measure: Count of Participants; unit: Participants
Arm/Group | Rituxan
Number analyzed (Participants) | 39
Participants | 32

2. Secondary Outcome: Number of Patients With Allograft Survival
Description: Graft survival in study participants
Time Frame: 12 months
Population: 32 patients were successfully transplanted during the study, of 39 total participants.
Measure: Count of Participants; unit: Participants
Arm/Group | Rituxan
Number analyzed (Participants) | 32
Participants | 28

3. Secondary Outcome: Reduction in Anti-HLA Antibodies
Description: Number of patients with a reduction in anti-HLA antibodies.
Time Frame: 9 months
Population: Donor specific antibodies (DSAs) assessed in transplanted population with DSA at time of transplant (32/39 patients transplanted during study, 23/32 with DSA at time of transplant)
Measure: Number; unit: percentage of patients
Arm/Group | Rituxan
Number analyzed (Participants) | 23
percentage of patients | 76

4. Secondary Outcome: Number of Acute Rejection Episodes
Description: Number of rejection episodes in study participants
Time Frame: 12 months
Population: 32 patients were successfully transplanted during the study, of 39 total participants. Only those who were transplanted were assessed for this endpoint.
Measure: Number; unit: rejection episodes
Arm/Group | Rituxan
Number analyzed (Participants) | 32
rejection episodes | 15

5. Secondary Outcome: Number of Patients Reporting a Serious Infection
Description: Infection rate in study participants
Time Frame: 12 months
Measure: Count of Participants; unit: Participants
Arm/Group | Rituxan
Number analyzed (Participants) | 39
Participants | 2

6. Secondary Outcome: Number of Adverse Events, Toxicity Assessments
Description: Adverse effects in study participants
Time Frame: 12 months
Measure: Number; unit: events
Arm/Group | Rituxan
Number analyzed (Participants) | 39
events | 14

ADVERSE EVENTS:
Time Frame: 1 year
Arm/Group | Rituxan
All-Cause Mortality (participants affected / at risk) | 3/39
Serious Adverse Events (participants affected / at risk) | 14/39
Other Adverse Events (participants affected / at risk) | 20/39
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Rituxan (N=39)
Fungal Infection (Infections and infestations) | 1 (1)
Parietal Cystic Lesion (Nervous system disorders) | 1 (1)
Bacterial Infection (Infections and infestations) | 1 (1)
Constipation (Gastrointestinal disorders) | 1 (1)
Urinary Incontinence (Renal and urinary disorders) | 1 (1)
Urinary Tract Obstruction (Renal and urinary disorders) | 1 (1)
Hyponatremia (Metabolism and nutrition disorders) | 1 (1)
Deep vein thrombosis (Vascular disorders) | 1 (1)
Cyst in Left Kidney (Renal and urinary disorders) | 1 (1)
Hematuria (Renal and urinary disorders) | 3 (3)
Hypertension (Cardiac disorders) | 1 (1)
Small Bowel Obstruction (Gastrointestinal disorders) | 1 (1)
Allograft Thrombosis (Renal and urinary disorders) | 1 (1)
Hemorrhagic Shock (General disorders) | 1 (1)
Fever (Nervous system disorders) | 1 (1)
Mild Hydronephrosis (Renal and urinary disorders) | 1 (1)
Gastritis (Gastrointestinal disorders) | 1 (1)
Coronary Artery Disease (Cardiac disorders) | 1 (1)
Bleeding from Incision Site (Surgical and medical procedures) | 1 (1)
OTHER ADVERSE EVENTS (reported when occurring in more than 3% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Rituxan (N=39)
Headache (Nervous system disorders) | 7 (7)
Urinary Tract Infection (Infections and infestations) | 2 (2)
Hypertension (Cardiac disorders) | 6 (6)
Hyperkalemia (Metabolism and nutrition disorders) | 4 (4)
Edema (Renal and urinary disorders) | 3 (3)
Cough (Respiratory, thoracic and mediastinal disorders) | 4 (4)
Itching (Skin and subcutaneous tissue disorders) | 5 (5)
Itchy or Sore Throat (Respiratory, thoracic and mediastinal disorders) | 4 (4)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2015-02-05): https://cdn.clinicaltrials.gov/large-docs/16/NCT01178216/Prot_SAP_000.pdf